CLINICAL TRIAL: NCT00639236
Title: Effectiveness and Safety of Inhaling Hypertonic Saline in the Functional Exercise Capacity of Patients With Chronic Obstructive Pulmonary Disease: a Randomized Trial
Brief Title: Effectiveness and Safety of Inhaling Hypertonic Saline in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Silvia Regina Valderramas, Evangelical Faculty of Paraná
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 017/04; 017/04
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Hypertonic saline; Quality of life; Dyspnoea.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: hypertonic saline — inhaled hypertonic saline (at a dose of 5 ml of a 3% solution) three times a week, combined with a program of physical exercises.

SUMMARY:
The use of inhaled hypertonic saline has been extensively documented in asthma, bronchiectasis, cystic fibrosis and COPD as method of bronchial challenge and sputum induction, but studies that evaluated others endpoints are required. The objective of this study was to analyse the effects of inhaling hypertonic saline compared with placebo with respect to functional exercise capacity, dyspnoea and quality of life. In a double-blind randomised parallel placebo-controlled trial, conducted at the Clínicas Integradas of the Evangelical Faculty of Paraná,sixty-eight patients (age 67 ± 6.5 years; FEV1 38.9 ± 16.2 predicted) were randomised to inhale 3% hypertonic saline (n=34) or placebo (n=34), combined with a program of exercise, three times a week, for 8-weeks.

DETAILED DESCRIPTION:
Background: The use of inhaled hypertonic saline has been extensively documented in asthma, bronchiectasis, cystic fibrosis and COPD as method of bronchial challenge and sputum induction, but studies that evaluated others endpoints are required. Objective: To analyse the effects of inhaling hypertonic saline compared with placebo with respect to functional exercise capacity, dyspnoea and quality of life. Design and Setting: This was a double-blind randomised parallel placebo-controlled trial, conducted at the Clínicas Integradas of the Evangelical Faculty of Paraná. Methods: sixty-eight patients (age 67 ± 6.5 years; FEV1 38.9 ± 16.2 predicted) were randomised to inhale 3% hypertonic saline (n=34) or placebo (n=34), combined with a program of exercise, three times a week, for 8-weeks. Results: After the 8-weeks the treatment period, both groups showed significant changes in functional exercise capacity (p<0,001), dyspnoea (p<0,001) and quality of life. When compared both groups, there was a significant improvement in placebo group in functional exercise capacity (p<0,001). Conclusion: the present study concluded that inhaling HS reduces the functional capacity, compared to placebo and being associated with the appearance of coughs and bronchial spasms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD diagnosis based on clinical findings and spirometry (FEV1 < 60% predict) according to American Thoracic Society20 clinically stable for at least the last month
* aged between 40 and 75 years old
* ex-smokers
* without severe and/or unstable heart disease or any other pathologic conditions that could impair physical activities (e.g., cerebrovascular diseases and rheumatism), were included.
* Respiratory medication was permitted, prior and throughout the duration of the study, such as bronchodilators and corticosteroids.

Exclusion Criteria:

* Patients with unstable lung disease (as evidenced by the administration of intravenous antibiotics for four weeks before screening)
* evidence of reactive airways (FEV1 ≥ 20 percent response to bronchodilatation or clinical diagnosis of asthma) were excluded

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-05; Primary Completion 2004-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | measured by the 6-minute walking distance (6MWD) test

SECONDARY OUTCOMES:
Dyspnoea | measured by the Medical Research Council dyspnoea score

CONTACTS AND LOCATIONS:
Overall Officials: Valderramas R Silvia, pHD, Principal Investigator — Federal University of São Paulo

REFERENCES:
- [Derived] Valderramas SR, Atallah AN. Effectiveness and safety of hypertonic saline inhalation combined with exercise training in patients with chronic obstructive pulmonary disease: a randomized trial. Respir Care. 2009 Mar;54(3):327-33. PMID 19245725